CLINICAL TRIAL: NCT07150637
Title: Development of an Early Warning Model for Intensive Care Unit-Acquired Weakness in Mechanically Ventilated Children: A Disease-Specific Cohort and Database Study
Status: Not yet recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: ICU-AW 20250824
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: ICU Acquired Weakness
Keywords: ICU acquired weakness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU-AW: Children receiving mechanical ventilation who developed ICU-AW at the study endpoint.
  Interventions: Diagnostic Test: ICU-AW
- without ICU-AW: Children receiving mechanical ventilation who did not developed ICU-AW at the study endpoint.

INTERVENTIONS:
Diagnostic Test: ICU-AW — The enrolled children receiving mechanical ventilation were grouped based on the occurrence of ICU-acquired weakness (ICU-AW) at the study endpoint.
  Groups: ICU-AW

SUMMARY:
Acquired weakness (AW) is a common complication among patients in the Intensive Care Unit (ICU). It is a systemic muscle weakness and dysfunction associated with critical illness, often related to prolonged bed rest, mechanical ventilation, systemic inflammatory response syndrome (SIRS), and multiple organ dysfunction syndrome (MODS). The primary clinical manifestations include weakness in limb and respiratory muscles, particularly diminished strength in distal muscle groups. As a result, the weaning process from mechanical ventilation becomes more challenging, leading to prolonged ICU stays, increased mortality, and a higher risk of long-term functional disability. The significance of AW lies not only in its substantial impediment to short-term recovery but also in its role as a core component of Post-Intensive Care Syndrome (PICS), profoundly affecting patients' long-term outcomes.

Mechanical ventilation is a vital life-support technology for critically ill children in the Pediatric Intensive Care Unit (PICU). However, complications associated with mechanical ventilation have garnered increasing attention, particularly Acquired Weakness in mechanically ventilated children. With improving survival rates in the PICU, a growing number of pediatric critical illness survivors are at risk of developing AW. Despite rapid advancements in pediatric critical care medicine in China, there is currently a lack of an early warning system for AW in children receiving mechanical ventilation, resulting in significantly delayed clinical interventions. This project aims to identify novel biomarkers for pediatric ICU-AW and develop an early warning model. It holds promise for transitioning from the traditional post-symptomatic diagnostic approach to subclinical prediction of AW in children, which is of great clinical value for reducing disability rates and optimizing critical care rehabilitation strategies.

DETAILED DESCRIPTION:
A prospective cohort study of mechanically ventilated children was established to systematically analyze epidemiological characteristics. The modified Pediatric Medical Research Council (MRC) muscle strength scale (pMRC) combined with simplified bedside neuroelectrophysiological testing (measurement of common peroneal nerve compound muscle action potential amplitude) was used to determine the occurrence rate, subtype distribution (CIP/CIM/Mixed), and natural disease course of intensive care unit-acquired weakness (ICU-AW) among mechanically ventilated children in China. An age-stratified model was applied to analyze differences in the occurrence rate of ICU-AW among children of different age groups. A Cox regression model was employed to quantify the dose-response relationship between dynamic parameters-such as duration of mechanical ventilation, cumulative doses of sedative and analgesic drugs, and glycemic variability-and the development of ICU-AW, and to construct a risk prediction nomogram.

Clinical parameters-including demographic characteristics, disease types, critical illness scores, treatment indicators such as mechanical ventilation parameters, laboratory indicators (e.g., inflammatory and biomarkers, metabolic genes), imaging data (muscle and diaphragmatic ultrasound, electrophysiology), molecular biomarkers, and muscle biopsy data-were integrated. Data mining and machine learning techniques were applied to develop an early warning model for ICU-AW based on Cox regression. A logistic regression preliminary screening model was constructed by integrating demographic characteristics and biomarkers. Quantitative parameters from muscle ultrasound (e.g., diaphragmatic excursion, muscle thickness) were incorporated, and dynamic risk assessment was optimized using the Random Forest algorithm. The sensitivity and specificity of the model were evaluated.

1. Study Design: This study employed a multicenter prospective cohort design.

1. Grouping: Pediatric patients undergoing mechanical ventilation were grouped based on the occurrence of ICU-AW at the study endpoint. The diagnostic criteria required meeting any one of the following: i) New-onset muscle dysfunction or weaning difficulty (unrelated to the primary disease, or in non-neuromuscular diseases with normal cardiopulmonary function); ii) Daily MRC score assessment for enrolled PICU patients [for patients under analgesic sedation, drug dosages were adjusted to maintain a modified Comfort-B sedation score between 11 and 23]. Patients with a total MRC score < 48 on two consecutive assessments 24 hours apart, and excluding those with other neuromuscular disorders, were assigned to the ICU-AW group; those with a total MRC score ≥ 48 were assigned to the non-ICU-AW group; patients who could not be evaluated were excluded. Subtype criteria: CIP: In addition to the above criteria, also meeting iii) Slowed sensory and/or motor nerve conduction velocity; CIM: In addition to criteria i and ii, also meeting iv) Reduced CMAP amplitude with prolonged duration, and normal SNAP amplitude; Mixed: Meeting both criteria iii and iv.
2. Sample Size Estimation (Data Management + Statistical Methods): The occurrence rate of pediatric ICU-AW was estimated at 2%. With a permissible error of 0.03 and a confidence level of 0.95, the sample size was calculated as 1500 cases using PASS software. Assuming a non-response rate of 10% among study subjects, the required sample size was N = 1500 / 0.9 = 1666 cases. Statistical analysis was performed using Stata 15.0 software. Continuous variables following a normal distribution in measurement data are presented as mean (SD); comparisons of means between groups were conducted using one-way and multi-way ANOVA. Those with a skewed distribution are presented as median (range or interquartile range, IQR). Count data (binary or multi-category) are expressed as incidence rates or composition ratios, with comparisons of incidence rates or composition ratios performed using the chi-square test. Logistic regression analysis was used to examine the relationship between biomarkers and the occurrence and development of ICU-AW, as well as the weight and contribution of each variable in the early warning model. ROC curve analysis was employed to assess model performance. A P-value < 0.01 was considered statistically significant for all analyses.

2. Case Collection and Data Analysis: An electronic database was established to collect clinical data from pediatric patients undergoing mechanical ventilation, including clinical baseline characteristics, laboratory test results, and imaging data. Each research center designated dedicated research personnel to begin enrolling study cases on the same start date (cases already hospitalized on the start date who met the inclusion criteria were enrolled). These personnel were responsible for data cleaning, organization, and standardization to ensure data quality. For all enrolled cases, demographic characteristics, clinical features, and laboratory test information were recorded in CRF forms on the day of enrollment (D0), day 3 (D3), day 10 (D10), the day of PICU discharge (Ddis), or the day of death (DD). Patient examinations for data collection were performed only when deemed appropriate by the physician. If an examination was not performed, the variable value was assumed to be normal or consistent with the previous measurement. Specific recorded information included:

1. Demographic characteristics: Age, sex, length/height, weight, body mass index.
2. Baseline clinical characteristics: Past medical history and underlying diseases, primary diagnosis upon PICU admission, critical illness score (PELOD-2), nutritional status (skinfold thickness/mid-upper arm circumference), CK, myoglobin, neurofilament light chain, a panel of twelve inflammatory factors, urinary titin, blood glucose, MRC muscle strength assessment, gastrocnemius muscle electrophysiology, rectus femoris muscle ultrasound, diaphragm thickness/excursion, treatments received (corticosteroids, e.g., dexamethasone, prednisone, methylprednisolone, hydrocortisone succinate; neuromuscular blocking agents, e.g., vecuronium), mechanical ventilation (duration in days, mode, fraction of inspired oxygen, mean airway pressure, tidal volume ml/kg, respiratory rate, P0.1), days on cardiopulmonary bypass (CPB), days on extracorporeal membrane oxygenation (ECMO), days of rehabilitation, whole-exome sequencing (WES) of family lineage, etc. Patient examinations for data collection were performed only when deemed appropriate by the physician. If an examination was not performed, the variable value was assumed to be normal or consistent with the previous measurement.
3. Determination of inflammatory markers: All inflammatory marker determinations were performed using EDTA-anticoagulated plasma samples. These included: Pro-inflammatory cytokines: IL-1β, IL-6, IL-8, TNF-α, IFN-γ, GM-CSF; Anti-inflammatory cytokines: IL-10, IL-13; Chemoattractant (CX3CL1), soluble intercellular adhesion molecule-1 (sICAM-1), soluble E-selectin (sE-selectin), and soluble P-selectin (sP-selectin). Each inflammatory marker was quantitatively determined using standardized immunoassay methods, such as ELISA (Enzyme-Linked Immunosorbent Assay).
4. Follow-up indicators: Nutritional status (skinfold thickness/mid-upper arm circumference), CK, myoglobin, blood glucose (D0, D3, D7, D10), MRC score, muscle ultrasound, diaphragm ultrasound, electromyography, muscle biopsy (if necessary) (D0, D3, D7, D10).
5. Outcome measures: The occurrence rate of ICU-AW in pediatric patients undergoing mechanical ventilation on day 3 or day 10. Defined as MRC score < 48, or slowed nerve conduction velocity on electromyography; CIP: Normal or mildly reduced nerve conduction velocity, reduced CMAP amplitude, reduced mixed SNAP amplitude; CIM: Normal or mildly reduced nerve conduction velocity, reduced CMAP amplitude, reduced muscle excitability to direct stimulation, increased CMAP duration, normal SNAP; or definitive diagnosis by muscle biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 28 days and 18 years;
2. Patients continuously admitted to the PICU during the study period and subjected to invasive mechanical ventilation.

Exclusion Criteria:

1. Mechanical ventilation duration < 72 hours;
2. Presence of primary central or neuromuscular diseases that significantly affect central or peripheral respiratory failure, including: traumatic brain injury, cerebrovascular disease history (e.g., cerebral hemorrhage, cerebral infarction), intracranial tumors, central nervous system infections, spinal cord injury, Guillain-Barré syndrome, porphyria, paraneoplastic neuropathy, etc.;
3. Conditions requiring immobilization such as limb joint surgery or fractures.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. Age between 28 days and 18 years;
  2. Patients continuously admitted to the PICU during the study period and subjected to invasive mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
The occurrence rate of ICU-AW | Diagnosis of ICU-AW in mechanically ventilated children was determined based on assessments at day 10.
  The occurrence rate of ICU-AW in mechanically ventilated children on day 10. ICU-AW was defined as: MRC score < 48, or slowed nerve conduction velocity on electromyography; CIP: normal or mildly reduced nerve conduction velocity, reduced CMAP amplitude, reduced mixed SNAP amplitude; CIM: normal or mildly reduced nerve conduction velocity, reduced CMAP amplitude, decreased muscle excitability to direct stimulation, increased CMAP duration, normal SNAP; or confirmed by muscle biopsy.

SECONDARY OUTCOMES:
Diaphragm Thickness: | mechanically ventilated children on day 0，day 3, day 7，day 10
  The thickness of the right hemidiaphragm was assessed using a linear array probe placed along the right midaxillary line at the 7th/8th and 8th/9th intercostal spaces. Under the 2D ultrasound mode, the imaging depth was appropriately adjusted to identify the target diaphragmatic region. The diaphragm appeared as a heterogeneous echogenic layer sandwiched between two hyperechoic lines representing the pleural and peritoneal layers. The distance between these two hyperechoic lines (excluding the thickness of the lines themselves) was measured as the diaphragm thickness.
Rectus Femoris Muscle Thickness and Cross-Sectional Area | mechanically ventilated children on day 0，day 3, day 7，day 10
  The thickness and cross-sectional area (CSA) of the rectus femoris muscle were assessed using a linear array transducer. The child was placed in the supine position with the knee extended. A generous amount of coupling gel was applied to minimize compression of the muscle by the transducer. The probe was positioned perpendicular to the long axis of the limb at the midpoint between the superior border of the patella and the anterior superior iliac spine. The rectus femoris muscle was identified, with its hyperechoic fascial layers serving as anatomical boundaries. Muscle thickness was defined as the distance between the superficial and deep fascial layers. The cross-sectional area was measured by tracing the circumference of the rectus femoris muscle along its fascial border.

CONTACTS AND LOCATIONS:
Locations (1):
- Children' hospital of Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kalb R. ICU-acquired weakness and recovery from critical illness. N Engl J Med. 2014 Jul 17;371(3):287. doi: 10.1056/NEJMc1406274. No abstract available. PMID 25014704
- [Background] Johnson RW, Ng KWP, Dietz AR, Hartman ME, Baty JD, Hasan N, Zaidman CM, Shoykhet M. Muscle atrophy in mechanically-ventilated critically ill children. PLoS One. 2018 Dec 19;13(12):e0207720. doi: 10.1371/journal.pone.0207720. eCollection 2018. PMID 30566470
- [Background] Zhang Z, Cai X, Ming M, Huang L, Liu C, Ren H, Qu D, Gao H, Cheng Y, Zhang F, Yang Z, Xu W, Miao H, Liu P, Liu Y, Lu G, Chen W. Incidence, outcome, and prognostic factors of prolonged mechanical ventilation among children in Chinese mainland: a multi-center survey. Front Pediatr. 2024 May 30;12:1413094. doi: 10.3389/fped.2024.1413094. eCollection 2024. PMID 38873585
- [Background] Zhang Z, Tao J, Cai X, Huang L, Liu C, Ren H, Qu D, Gao H, Cheng Y, Zhang F, Yang Z, Xu W, Miao H, Liu P, Liu Y, Lu G, Chen W. Clinical characteristics and outcomes of children with prolonged mechanical ventilation in PICUs in mainland China: A national survey. Pediatr Pulmonol. 2023 May;58(5):1401-1410. doi: 10.1002/ppul.26332. Epub 2023 Feb 8. PMID 36705329
- [Background] Banwell BL, Mildner RJ, Hassall AC, Becker LE, Vajsar J, Shemie SD. Muscle weakness in critically ill children. Neurology. 2003 Dec 23;61(12):1779-82. doi: 10.1212/01.wnl.0000098886.90030.67. PMID 14694046